CLINICAL TRIAL: NCT03204721
Title: Prevention of Graft-versus-host Disease in Patients Treated With Allogeneic Stem Cell Transplantation: Possible Role of Extracorporeal Photophoresis
Brief Title: Prevention of GVHD in Patients Treated With Allogeneic SCT: Possible Role of Extracorporeal Photophoresis
Acronym: GVHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Tobias Gedde-Dahl d.y., Consultant hematologist MD,PhD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2016/1130
Record Dates: First submitted 2017-06-01; First posted 2017-07-02 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Graft-Versus-Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — Photopheresis

STUDY DESIGN:
Intervention Model Description: Patients admitted for allogeneic stamcelltransplantation who consent participation in the study are randomized 1:1, either to receive ECP or no-ECP
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extracorporeal photophoresis (Active Comparator): The treatment procedure of ECP consists of three steps. First, the leukocytes are removed by apheresis; second, the mononuclear cells are primed with the photosensitizing agent 8-methoxypsoralen; then third, these cells are exposed to radiation with ultraviolet A light before they are re-infused into the patient.
  Interventions: Other: Extracorporeal photophoresis (ECP)
- Controll (No Intervention): No procedure

INTERVENTIONS:
Other: Extracorporeal photophoresis (ECP) — The treatment procedure of ECP consists of three steps. First, the leukocytes are removed by apheresis; second, the mononuclear cells are primed with the photosensitizing agent 8-methoxypsoralen; then third, these cells are exposed to radiation with ultraviolet A light before they are re-infused into the patient
  Arms: Extracorporeal photophoresis

SUMMARY:
The main aim is to test the preventive use of extracorporeal photophoresis (ECP) against development of graft-versus-host disease (GVHD) in patients undergoing allogeneic stem cell transplantation for hematological malignancy.

DETAILED DESCRIPTION:
Allogeneic stem cell transplantation represents the only available long-term control and possible cure of a number of hematological malignancies. A major obstacle to this treatment is the development of graft-versus-host disease (GVHD), affecting the majority of transplanted patients to some extent. Today, combinations of various cytotoxic and immunosuppressive drugs are used to prevent and treat GVHD, but many of them are associated with severe side-effects. Extracorporeal photophoresis (ECP) offers an alternative to chemo- and immunosuppressive therapy and confers apparently only mild side effects. The postulated rationale of ECP is to treat the patient's white blood cells ex vivo with ultraviolet irradiation after sensitization with 8-methoxypsoralen to dampen their immunoactivity. After engraftment the intervention group receives 2 consecutive ECP every week in 2 weeks then 1 ECP every week in 4 weeks ( a total of 8 ECP procedures).

ELIGIBILITY:
Inclusion Criteria:

* Provide written consent to participate
* Understand Norwegian or English
* No previous history of malignant disease
* No contraindication to ECP-treatment or undergone previous ECP treatment

Exclusion Criteria:

* (in addition to those regarding eligibility for transplantation itself):

  * Unwilling to provide written consent to participate
  * Unable to cooperate as judged by the responsible physician
  * ECOG status > 2 at time of inclusion
  * Using anti-inflammatory or cytotoxic drugs other than those that are part of the treatment of the current hematological malignancy
  * Known allergy to psoralens or citrate products
  * Splenectomy
  * Pregnancy/lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2017-06-21 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Reduce the frequency of GVHD by preventive treatment with ECP of patients undergoing allogeneic stem cell transplantation for hematological malignancies | up to 1 year after allogeneic stamcell transplantation
  GVHD is measured according to internationally recognized criteria

SECONDARY OUTCOMES:
Number of survivors the first year after transplantation | Through study completion, and until 1 year after study start
  In the follow-up periode mortality rate in both groups is registered
Number of patients who relapsed the first year after transplantation Number of patients who relapsed the first year after transplantation Number of patients who relapsed the first year after transplantation | Through study completion, and until 1 year after study start
  In the follow-up periode relapse rate in both groups is registered
Quality of life (QoL) the first year after transplantation | Through study completion, and until 1 year after study start
  In the follow-up periode EORTC-QLQ-C30 scores in both groups are registered
Assessment of vitamin A derivatives | From randomization to 3 months after transplantation
  Measurement of retinoids and carotenoids in plasma before and after ECP treatment
Determination of microbiota | Through study completion, and until 1 year after study start
  Assaying fecal microbiota from both study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Geir E Tjønnfjord, Prof,MD,PhD, Study Chair — Oslo University Hospital HF, Department of Haematology Rikshospitalet; Per Ole Iversen, Prof,MD,PhD, Study Chair — Oslo University Hospital HF, Department of Haematology Rikshospitalet
Locations (1):
- Tobias Gedde-Dhl, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No